CLINICAL TRIAL: NCT06314542
Title: Quantitative Evaluation of the Impact of Relaxing Eligibility Criteria on the Risk-benefit Profile of Drugs for Lung Cancer Based on Real-world Data
Brief Title: Quantitative Evaluation of the Impact of Relaxing Eligibility Criteria for Lung Cancer Based on Real-world Data
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: REC-001
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: relaxing eligibility criteria — Quantitative evaluation of the impact of relaxing eligibility criteria on the risk-benefit profile of drugs for lung cancer based on real-world data

SUMMARY:
Eligibility criteria for cancer drug trials are generally too stringent, leading to key issues such as low enrolment rates and lack of population diversity. In order to evaluate the REC of NSCLC drug trials, this study will use deep learning methods to construct a structured real-world database of NSCLC across dimensions, and quantitatively assess the independent contribution of changes in each eligibility criterion to patient numbers, clinical efficacy and safety.

DETAILED DESCRIPTION:
Restrictive eligibility criteria in cancer drug trials result in low enrollment rates and limited population diversity. Relaxed eligibility criteria (REC) based on solid evidence is becoming necessary for stakeholders worldwide. However, the absence of high-quality, favorable evidence remains a major challenge. This study presents a protocol to quantitatively evaluate the impact of relaxing eligibility criteria in common non-small cell lung cancer (NSCLC) protocols in China, on the risk-benefit profile. This involves a detailed explanation of the rationale, framework, and design of REC.

To evaluate our REC in NSCLC drug trials, we will first construct a structured, cross-dimensional real-world NSCLC database using deep learning methods. We will then establish randomized virtual cohorts and perform benefit-risk assessment using Monte Carlo simulation and propensity matching. Shapley value will be utilized to quantitatively measure the effect of the change of each eligibility criterion on patient volume, clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

Patients in the database were considered to be part of the real-world cohort if they were (1) diagnosed with NSCLC according to the tenth revision of the international classification of diseases (ICD-10) code; (2) diagnosed with stage IIIB, IIIC, IV NSCLC between 1 January 2013 and 31 December, 2022; (3) had at least two documented clinical visits on or after 1 January 2013.

Exclusion Criteria:

（1）NSCLC in stage I-IIIa

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Those patients diagnosed with primary NSCLC in stage IIIb-IV, are the study population.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Scale of eligibility criteria | 2024.12.31
  Lung cancer clinical trial protocol eligibility criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, doctor, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China